CLINICAL TRIAL: NCT07100223
Title: Awareness-Based Parentıng And Bırth Preparatıon Educatıon Gıven To Couples; Impact Of Maternal-Paternal Attachment, Bırth Parameters And Postpartum Rapport
Brief Title: Awareness-Based Parentıng And Bırth Preparatıon Educatıon Gıven To Couples
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, MERVE GÜL TİREN, specialist nurse, Kayseri Training and Research Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: KayseriTRH
Record Dates: First submitted 2024-05-15; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Educational Problems
Keywords: ADAPTATION; ATTACHMENT; MINDFULNESS; PARENT
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: An experimental design with pretest posttest control group will be used.
Who Masked: Participant
Masking Description: In the study, couples will be assigned to groups according to the randomization list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION GROUP (Experimental): 15 couples who meet the inclusion criteria will be assigned to groups according to the parental randomization list. Awareness-Based Parenting and Birth Preparation Training will be given as group training on Mondays of each week, during the hours when the pregnancy school does not provide training.
  Interventions: Other: EDUCATION
- CONTROL GROUP (Experimental): No intervention will be made to the parents in the control group other than the birth preparation training carried out by Kayseri City Hospital.
  Interventions: Other: EDUCATION

INTERVENTIONS:
Other: EDUCATION — Assignment to the intervention and control groups will be made by randomization method.
  Before training is given to the intervention and control groups, Parental Introduction Form, Conscious Awareness Scale, Prenatal Attachment Scale, Prenatal Attachment Scale, Fathers' Fear of Birth Scale, Wijma Birth Expectation/Experience Scale Version A will be applied.
  After parents attend a 1-week birth preparation training at Kayseri City Hospital Pregnancy School, they will participate in a 9-week Awareness-Based Parenting and Birth Preparation Training.
  After the training is completed; Conscious Awareness Scale, Prenatal Attachment Scale, Prenatal Attachment Scale, Fathers' Fear of Birth Scale, Wijma Birth Expectation/Experience Scale Version A will be applied.
  Wijma Birth Expectation/Experience Scale Version B will be administered to mothers on the 1st postpartum day.

SUMMARY:
One of the behavioral intervention programs used to adapt to the changes experienced during pregnancy, birth and postpartum and to maintain a healthy transition to parenthood is Conscious Awareness-Based Practices Conscious awareness is an experiential process in which attention is directed purposefully and consciously to what is happening in the body and mind at that moment, and the content that emerges as a result of these observations is accepted with curiosity, understanding and compassion, without being judged, analyzed, or reacted . Due to their stated effects, these interventions help parents improve their awareness and acceptance of thoughts, feelings, and body sensations, reduce reactivity, avoid disturbing experiences, accept the roles and responsibilities of parenting in a non-judgmental manner, learn to use mechanisms to cope with the stress of parenting, and help themselves and the child. It is important to enable people to show compassion .

Awareness-based training can be integrated into birth preparation training as it is a method that can be used to improve birth parameters.

Awareness-Based Parenting and Birth Preparation Training applied during the transition to parenthood is important as it will increase the quality of pregnancy, birth and postpartum care, as it will increase competence and adaptation to parenting roles, facilitate the birth process, and ensure maternal and paternal attachment. For all these reasons, this research was planned to investigate the effects of Awareness-Based Parenting and Birth Preparation Training given to couples on maternal-paternal attachment, birth parameters and postpartum adaptation. It is thought that the training that parents receive to be aware of their own body and birth process will make a positive contribution to pregnancy, birth and the postpartum process.

DETAILED DESCRIPTION:
One of the behavioral intervention programs used to adapt to the changes experienced during pregnancy, birth and postpartum and to maintain a healthy transition to parenthood is Conscious Awareness-Based Practices .Conscious awareness is an experiential process in which attention is directed purposefully and consciously to what is happening in the body and mind at that moment, and the content that emerges as a result of these observations is accepted with curiosity, understanding and compassion, without being judged, analyzed, or reacted.Due to their stated effects, these interventions help parents improve their awareness and acceptance of thoughts, feelings, and body sensations, reduce reactivity, avoid disturbing experiences, accept the roles and responsibilities of parenting in a non-judgmental manner, learn to use mechanisms to cope with the stress of parenting, and help themselves and the child. It is important to enable people to show compassion .

Awareness-based training can be integrated into birth preparation training as it is a method that can be used to improve birth parameters.

The word parent means mother and father according to the Turkish Language Association. It is also described as a nuclear family and represents a child's mother and father. The meaning of being a parent is defined as constantly providing care, needs and support for a child for development and survival .

Becoming a parent is one of the developmental transition periods that adds new roles and responsibilities to an individual's life and involves radical changes .This process of change is called the transition period to parenthood .Although there are many different opinions about when the transition to parenthood begins and ends, the most widely accepted view is that it begins with pregnancy in individuals who become mothers/fathers for the first time and ends within a few months after birth. The transition period is followed by the parenthood period .

The transition to parenthood also brings about parent-infant bonding. The term attachment refers to the ability to establish and maintain an emotionally positive, reciprocal, helpful relationship between infants and parents. If the relationship is properly established, adults adapt themselves to their babies, and babies give adults clues about their needs. This relationship, which develops in the early period, has an important place in the physical, psychological and intellectual development of the child and continues its effectiveness throughout life. The family-infant attachment process develops in three periods: pregnancy, birth and postpartum .During pregnancy, it is important for parents to feel and caress their baby physically, to believe that their baby is establishing a relationship with them, to talk to the fetus, to say its name, to think about their baby, to feel positive emotions about their baby, and to imagine their baby's future situation for the development of attachment.. It is stated that the attachment that begins during pregnancy gradually increases as pregnancy progresses and becomes stronger after the baby is born.In a study examining attachment, it was determined that there was a strong and significant relationship between prenatal attachment and postpartum attachment .Since the aware emotions created by attachment are motivating during pregnancy and facilitate adaptation to the parenting role, they also positively affect the parent-infant adaptation process.

Pregnancy is seen as an important preparation period for parenthood in which physiological, psychological, social and emotional changes occur and requires adaptation to these changes. Especially individuals who will be mothers and fathers for the first time may experience a feeling of uncertainty regarding the process of pregnancy, birth and the changes experienced in the postpartum period. Parents want the pregnancy process to be smooth and the birth to be painless and with high satisfaction.However, in this process, they experience complex emotions such as anxiety, fear and excitement together. Fears generally arise from episiotomy during vaginal birth, the thought that there may be a tear in the perineum, the pain that will be felt during all these processes, and the responsibilities of baby care that come with being a parent .

There are many training programs on attitudes and behaviors towards parents in order to facilitate individuals' adaptation to these changes and to better manage their transition to parenthood. These programs have a positive effect on the individual well-being of parents, their ability to acquire parenting skills in a healthy way, and the healthy development of the child. By supporting the uncertainty in this transition process with educational programs in the prenatal period, family-infant bonding and adaptation can be achieved, and pregnancy, birth and the postpartum process can be continued in a healthy way .

One of the behavioral intervention programs used to adapt to the changes experienced during pregnancy, birth and postpartum and to maintain a healthy transition to parenthood is Conscious Awareness-Based Practices. Conscious awareness is an experiential process in which attention is directed purposefully and consciously to what is happening in the body and mind at that moment, and the content that emerges as a result of these observations is accepted with curiosity, understanding and compassion, without being judged, analyzed, or reacted. It is a skill that allows us not to be passive towards everything that is happening right now, and it is associated with all our positive, negative and neutral experiences, reducing all levels of suffering and increasing our state of well-being . Due to their stated effects, these interventions help parents improve their awareness and acceptance of thoughts, feelings, and body sensations, reduce reactivity, avoid disturbing experiences, accept the roles and responsibilities of parenting in a non-judgmental manner, learn to use mechanisms to cope with the stress of parenting, and help themselves and the child. It is important to enable people to show compassion.

In a study conducted in Turkey, a conscious awareness-based approach was applied to women who were followed up in a clinic with a diagnosis of premature rupture of membranes, and its effect on their adaptation to motherhood in the prenatal period, maternal attachment levels, and adaptation to motherhood in the postpartum period was evaluated. It was determined that after the intervention, there was an increase in women's competence levels regarding pregnancy acceptance, birth preparation, maternal attachment and the maternal role . In a study that conducted a systematic review of mindfulness-based interventions during pregnancy, it was found that it was useful for overcoming undesirable situations such as anxiety, depression, fear of birth and perceived distress and increased psychological well-being. As a result of the study conducted to increase birth self-efficacy; Awareness and birth self-efficacy levels increased significantly. ) emphasized that mindfulness interventions implemented to improve maternal outcomes have positive effects on maternal well-being. They reported that this state of well-being not only psychologically but also physically regulates blood pressure and blood sugar, slows down heart rate, and improves fatigue and activity levels.

Awareness-based training can be integrated into birth preparation training as it is a method that can be used to improve birth parameters. When the literature is examined, although there are studies examining the effects of Awareness-Based Parenting and Birth Preparation Education on mothers in the perinatal period, studies in which fathers are included in the application and studies examining the relationship between adaptation and attachment and awareness are limited. It is stated that actively involving both parents in group-based parenting training is more effective in increasing the efficiency of the program stated that conscious awareness is an important feature of transition. The higher the individual's awareness of the new role he will assume at the end of the transition, the higher his level of competence and success in the role will be Therefore, Awareness-Based Parenting and Birth Preparation Training, applied during the transition to parenthood, is important as it will increase the quality of pregnancy, birth and postnatal care, as it will increase competence and adaptation to parenting roles, facilitate the birth process, and ensure maternal and paternal attachment. For all these reasons, this research was planned to investigate the effects of Awareness-Based Parenting and Birth Preparation Training given to couples on maternal-paternal attachment, birth parameters and postpartum adaptation. It is thought that the training that parents receive to be aware of their own body and birth process will make a positive contribution to pregnancy, birth and the postpartum process.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 18-35 age group,
* First pregnancy,
* 24-28. week of pregnancy,
* Those who applied to the Pregnancy Polyclinic between the dates of the research and were accepted to the Pregnancy School training,
* At least literate education level,
* People who are open to communication will be included in the study.

Exclusion Criteria:

* Those with psychiatric disorders,
* Pregnant women with pregnancy-related risk factors that may lead to premature birth,
* Pregnant women with chronic diseases that may lead to the risk of premature birth will be excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participation of both parents in birth preparation training will be ensured.
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
1. Mindful Attention Awareness Scale(MAAS) total score to assess change in trait mindfulness | [Time Frame: Baseline (pre-intervention) and post-intervention (week 8)]
  The MAAS is a 15-item self-report questionnaire developed by Brown & Ryan (2003) and adapted into Turkish by Özyeşil et al. (2011). It measures the frequency of mindful states in daily life using a 6-point Likert scale (1 = Almost always to 6 = Almost never), with total scores ranging between 15 and 90. Higher scores reflect higher dispositional mindfulness.
  Unit of Measure:
  Total Score (15-90)

SECONDARY OUTCOMES:
2. Wijma Delivery Expectancy Questionnaire (W-DEQ)total score to assess fear of childbirth | [Time Frame: Baseline (gestational week 28-30) and post-intervention (gestational week 36)
  The W-DEQ is a 33-item self-report questionnaire developed by Wijma et al. (1998) to assess fear of childbirth. Items are scored on a 6-point Likert scale (0 = Not at all to 5 = Extremely), with total scores ranging from 0 to 165. Higher scores indicate greater fear. The Turkish version has been validated in pregnant populations.
  Unit of Measure:
  Total Score (range: 0-165)
3. Visual Analog Scale (VAS)score to assess perceived labor pain | [Time Frame: IMMEDIATELY AFTER BIRTH]
  Pain intensity will be measured using the Visual Analog Scale (VAS), a self-reported measure where participants rate their pain on a scale from 0 (no pain) to 10 (worst imaginable pain). The score reflects the subjective intensity of labor pain during active labor. VAS is a widely used and validated tool for assessing acute pain.
  Unit of Measure:
  Score (range: 0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Kocasi̇nan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meleis, A. I. (2010). Transitions theory: Middle range and situation specific theories in nursing research and practice. Springer publishing company. Muller, M.E. (1994). A questionnaire to measure mother- to- infant attachment, J Nurs Meas, 2(2), 129-41. Onat, G. (2021). Farkındalıkla Emzirme Süt Arttırma ve Doğum. Akademisyen Kitabevi. Özyeşil, Z., Arslan, C., Kesici, Ş., Deniz, M.E. (2011) Bilinçli farkındalık ölçeğini Türkçeye uyarlama çalışması. Eğitim ve Bilim Dergisi, 36(160), 224-35. Pallant, J. (2020). SPSS hayatta kalma kılavuzu: IBM SPSS kullanarak veri analizine yönelik adım adım bir kılavuz . McGraw-hill eğitimi (İngiltere). Pan, W.L., Chang, C.W., Chen, S.M., & Gau, M.L. (2019a). Assessing the effectiveness of mindfulness-based programs on mental health during pregnancy and early motherhood-a randomized control trial. BMC Pregnancy and Childbirth, 19(1), 1-8. doi: 10.1186/s12884-019-2503-4 Prinds, C., Hvidtjørn, D., Skytthe, A. (2016). Danimarkalı ilk kez anne olanlar arasında dua ve meditasyon - bir anket çalışması. BMC Gebelik Doğum 16, 8. https://doi.org/10.1186/s12884-016-0802-6 Schumacher, K. L., Meleis, A. L. (1994). Transitions: A central concept in nursing. Image: The Journal of Nursing Scholarship, 26(2), 119-127 Seyhan A.G. (2023). Birlikte Ebeveynliğe Geçiş Programı'nın (Begep) Birlikte Ebeveynlik Algıları Üzerindeki Etkisi. Yüksek Lisans Tezi, Aydın. Shorey, S., Ang, L., Yin, C. A. (2019). Systematic mixed-studies review on mindfulness-based childbirth education programs and maternal outcomes. Nursing Outlook, 67(6), 696-706. Sluijs, A.M., Wijma, K., Cleiren, M.P., Van Lith, J.M., Wijma, B. (2020). Preferred and actual mode of delivery in relation to fear of childbirth. Journal of Psychosomatic Obstetrics & Gynecology, 1-9. Şatır, D. G., Kavlak, O. (2021). Validity and reliability of Turkish version of "Paternal Antenatal Attachment Questionnaire":"Paternal Antenatal Bağlanma Ölçeği" nin Türkçe versiyonunun geçerlik ve güvenirlik çalışması. Journal of Human Sciences, 18(1), 1-11. Taşçı, K., Samiye, Mete. (2010). Postpartum Kendini Değerlendirme Ölçeğinin Geçerlik Ve Güvenirlik Çalışması. Anadolu Hemşirelik Ve Sağlık Bilimleri Dergisi, 10(2), 20-29. Taşkın L. (2020). Doğum ve Kadın Sağlığı Hemşireliği. 16. Baskı, Ankara, Akademi Yayınevi, 157-184. Türk Dil Kurumu (TDK) Sözlükleri.(2023). https://sozluk.gov.tr/ Uçar, E., Beji, D.N.K. (2013) Wijma Doğum Beklentisi/Deneyimi Ölçeği B Versiyonu'nun Geçerlik Ve Güvenirlik Çalışması.Yüksek Lisans Tezi. İstanbul. Van Vreeswijk, M., Broersen, J., Schurink, G. (2014). Mindfulness and Schema Therapy: A Practical Guide. Veringa, I.K., Bruin, E.I., Bardacke, N. (2016). I've changed my mind', Mindfulnessbased childbirth and parenting (MBCP) for pregnant women with a high level of fear of childbirth and their partners: study protocol of the quasi-experimental controlled trial. BMC Psychiatry, 16, 377. Vieten, C., Astin, J. (2008). Effects of a mindfulness-based intervention during pregnancy on prenatal stres and mood: results of a pilot study. Archives of Womens' Mental Health, 11(1), 67-74. Vreeswijk, M. V., Broersen, J., Schurink, G. (2019). Mindfulness ve Şema Terapi Uygulama Rehberi. İstanbul: Psikonet Yayıncılık. Vural Batık, M., Kalkan, M. (2018). Ebeveyn Adayları İçin Evlilik Okulu Psikolojik Danışman El Kitabı, Anı Yayınları. Wijma, K., Wijma, B., Zar, M. (1998). Psychosomatic aspects of W-DEQ: A new questionnaire for measurement of fear of childbirth, Journal of Psychosomatic Obstetric Gynaecology, 19(4), 84-97 Xiao, X., Loke, A.Y. (2022). Intergenerational co-parenting in the postpartum period: A concept analysis. Midwifery, 107, 103275. Yılmaz, S. D.(2013). Prenatal anne-bebek bağlanması. Hemşirelikte Eğitim ve Araştırma Dergisi, 10(3), 28-33. Young, C., Roberts, R., Ward, L. (2020). Enhancing resilience in the transition to parenthood: a thematic analysis of parents' perspectives. Journal of Reproductive and Infant Psychology, 39(4), 358-370.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT07100223/Prot_SAP_000.pdf